CLINICAL TRIAL: NCT01925443
Title: Effects of Low Power Laser Therapy on Muscle Performance Isokinetic Pre-exercise in Individuals With Diabetes Mellitus Type II
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: technical problems with equipment from the main outcome
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Cid André Fidelis de Paula Gomes, Professor, University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1146-7109
Record Dates: First submitted 2013-06-08; First posted 2013-08-19 (Estimated); Last update posted 2015-12-03 (Estimated); Status verified 2015-12

CONDITIONS: Diabetes Mellitus Non-insulin-dependent
Keywords: diabetes mellitus non-insulin-dependent; low level laser therapy
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Low-Level Light Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- low level laser therapy (Experimental): individuals will be subject to the application of low level laser therapy, but this group will have three subdivisions related to dose in joules that will be administered to the individual, and J 4, J 6, 8 J. To be administered in the quadriceps muscle.
  Interventions: Other: Low level laser therapy
- Control Group (No Intervention): will consist of individuals diagnosed with diabetes mellitus non-insulin-dependent, however, will not perform low level laser therapy, participate only in the evaluations
- Placebo group (Experimental): individuals will be subject to the application of low level laser therapy but with a dose of 0 Joules.
  Interventions: Other: Low level laser therapy

INTERVENTIONS:
Other: Low level laser therapy — Will be performed irradiation with low-intensity laser in quadriceps muscle
  Arms: Placebo group; low level laser therapy

SUMMARY:
The low level laser therapy is able to improve immediately and long term (after 4 weeks of treatment, 3 days per week resulting in 12 applications of low level laser therapy) isokinetic muscle performance of the quadriceps femoris muscle (peak torque, total muscular work , maximum power and fatigue index - normalized by body weight) pre-exercise concentric isokinetic quadriceps femoris muscle in subjects with diabetes mellitus non-insulin-dependent.

DETAILED DESCRIPTION:
The low level laser therapy is able to improve after 4 weeks of treatment, 3 days per week resulting in 12 applications of low level laser therapy, the indicators: The low level laser therapy is able to improve immediately and long term (after 4 weeks of treatment, 3 days per week resulting in 12 applications of low level laser therapy), the indirect blood markers for muscle damage that evaluate the enzymatic activity of creatine Kinase (CK) and Lactate Dehydrogenase (LDH) and the visual analog scale (VAS-F) for fatigue, improves indicators F 2.2 point of the WHOQOL-100 for fatigue, improvement in functional indicators of the lower lower Extremity functional regarding Scale, functional improvement in performance in the execution of the test stand and sit and walk test six minutes, the indicators for quality improvement of life questionnaire for the Diabetes Quality of Life Measure and emotional states through the questionnaire Problems Areas in Diabetes Scale. Eligibility criteria: Diagnosis for Diabetes mellitus non-insulin-dependent confirmed by the individual physician, presenting between 30 to 70 years.Exclusion criteria: Diagnosis of cardiovascular disorders, diagnosis of diabetic neuropathy, which have a skin lesion or local infection (quadriceps), history of musculoskeletal injuries in the last 6 months or during the study, individuals unable to perform the assessment protocols / exercise so satisfactory, those who are doing some kind of regular physical activity and who underwent alcohol intake in the 24 hours before any of the stages of the study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis for Diabetes mellitus non-insulin-dependent
* Age between 30 to 70 years

Exclusion Criteria:

* Diagnosis of cardiovascular disorders
* Diagnosis of diabetic neuropathy,
* Skin lesion or local infection (quadriceps)
* History of musculoskeletal injuries in the last 6 months or during the study
* Individuals unable to perform the assessment protocols or exercise
* Regular physical activity
* Underwent alcohol intake in the 24 hours before any of the stages of the study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2015-12; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Muscle function | 2 Years
  Will use the isokinetic dynamometer to test and evaluate the human musculoskeletal system: peak torque and muscle fatigue of quadriceps.

SECONDARY OUTCOMES:
Muscle damage | 2 year
  Will be evaluated blood markers (creatine kinase and lactate dehydrogenase) as indirect markers of muscle damage by spectrophotometry using kits specific reagents.
Muscle fatigue | 2 years
  In order to assess self-perceived fatigue in day-to-day and immediately after the fatigue protocol will be used two instruments: a visual analog scale (VAS-F) and the question of F2.2 instrument for assessing quality of life World Health Organization (WHOQOL-100).
Functionality | 2 years
  Functionality will be evaluated using the following assessment tools: Stand and sit test, Six-minute walk test, and Lower Extremity Functional Scale.
Quality of life | 2 years
  The quality of life will be assessed by the questionnaire "Diabetes Quality of Life Measure"

CONTACTS AND LOCATIONS:
Overall Officials: Cid Gomes, MSc, Principal Investigator — University of Nove de Julho
Locations (1):
- University of Nove de Julho, São Paulo, São Paulo, Brazil

REFERENCES:
- See also: Related Info — http://www.uninove.br